CLINICAL TRIAL: NCT00361439
Title: Treatment of Olfactory Dysfunction in Seasonal Allergic Rhinitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped early due to slow accrual.
Sponsor: University of Chicago (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14757A (P04908); IRB #14757A
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone (Active Comparator): Mometasone intranasal steroid therapy daily for 2 weeks
  Interventions: Drug: Mometasone
- Placebo (Placebo Comparator): 2 puffs of placebo spray in each nostril once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone — 2 puffs in each nostril once daily of nasal spray
  Other Names: Nasonex
  Arms: Mometasone
Drug: Placebo — 2 puffs in each nostril once daily of nasal spray
  Arms: Placebo

SUMMARY:
People with allergies frequently complain of a loss or reduction in the sense of smell.

In this study, the investigators propose to perform a randomized, double blind, placebo controlled parallel study of subjects with nasal allergies and decreased smell to determine the effect of a treatment for allergies on the sense of smell.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 59 years of age.
2. Seasonal allergic rhinitis by clinical history, with symptoms of impaired olfaction.
3. Positive skin or RAST test to allergen.
4. Symptoms of olfactory dysfunction.
5. No significant history of chronic sinusitis.

Exclusion Criteria:

1. Women of childbearing potential not using the contraception method(s) (Birth control pills, depo Provera, double barrier) as well as women who are breastfeeding.
2. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (heart, lung, kidney, neurological, oncologic or liver disease).
3. Use of any other investigational agent in the last 30 days.
4. Absence of olfactory or nasal symptoms.
5. Use of medications that may affect olfaction.
6. Medical conditions that may affect olfaction.
7. Smoking.
8. URI at the time of screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayant M Pinto, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Sivam A, Jeswani S, Reder L, Wang J, DeTineo M, Taxy J, Baroody FM, Naclerio RM, Pinto JM. Olfactory cleft inflammation is present in seasonal allergic rhinitis and is reduced with intranasal steroids. Am J Rhinol Allergy. 2010 Jul-Aug;24(4):286-90. doi: 10.2500/ajra.2010.24.3478. PMID 20819468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled during relevant allergy seasons in Chicago, IL, from 2006 to 2008.
Groups:
- Mometasone: Active intranasal steroid therapy daily for 2 weeks
- Placebo: 2 puffs of placebo spray once daily
Period: Overall Study
Arm/Group | Mometasone | Placebo
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 40 [24 to 49] | 38 [23 to 52] | 39 [23 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
Allergen sensitivity [Number; unit: participants]
  Ragweed | 5 | 6 | 11
  Grass | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Histological Findings
Description: Number of eosinophils per high-powered field (HPF) in olfactory biopsy taken after 2 weeks of study treatment (higher values indicate greater inflammation); average of three HPF reported
Time Frame: 2 weeks
Measure: Median (Full Range); unit: eosinophils per HPF
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 8 | 9
eosinophils per HPF | 0.167 [0 to 1.33] | 2.67 [1.33 to 11]
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other; p < 0.02, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score at 2 Weeks
Description: A decrease in scores between visits signifies an improvement in nasal symptoms. The total nasal symptom score can range from 0 to 27.
Time Frame: baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | -12 [-18 to -2] | -5 [-13 to 13]
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other; p < 0.023, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Nasal Peak Inspiratory Flow at 2 Weeks
Description: An increase between visits indicates improved nasal airflow.
Time Frame: baseline and 2 weeks
Measure: Median (Full Range); unit: liters per minute
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 8 | 9
liters per minute | 19.2 [-3.3 to 56.7] | -37.5 [-58 to 5]
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other; p < 0.002, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Percentage of Eosinophils at 2 Weeks
Description: A decrease between visits signifies a reduction in inflammation.
  Calculated from cytology specimens obtained by lavage.
Time Frame: baseline and 2 weeks
Measure: Median (Full Range); unit: percentage of eosinophils
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 8 | 9
percentage of eosinophils | -1.35 [-12.9 to 4.2] | -0.1 [-53.9 to 0.8]
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other; p < 0.010, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the two weeks of treatment
Arm/Group | Mometasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes